CLINICAL TRIAL: NCT07339449
Title: Intraoperative Multimodal Monitoring as a Means in Reducing the Duration of Mechanical Ventilation in High-Risk Patients Undergoing Major Abdominal Procedures - A Pilot Study
Acronym: IMMEDIUM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Dubrava (Other)
Responsible Party: Principal Investigator, Jasminka Persec, MD, PhD, Intraoperative multimodal monitoring as a means in reducing the duration of mechanical ventilation in high-risk patients undergoing major abdominal procedures - a pilot study, University Hospital Dubrava
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2025/ 0603-8
Record Dates: First submitted 2026-01-13; First posted 2026-01-14 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Major Abdominal Surgeries; Mechanical Ventilation
Keywords: Abdominal surgery; minimally invasive; cardiac output; cerebral oximetry; multimodal monitoring

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Interventional (Experimental): Radial artery cannulation insertion before induction, LiDCOrapid®, Rainbow®, and haemoglobin attachment to the Root® monitor. Baseline measurements of MAP and CO, DO2 will be calculated from CO and haemoglobin values. SedLine® and O3® sensors will be placed to measure baseline anaesthetic depth and rSO2 before pre-oxygenation. Noradrenaline infusion will be initiated.Anaesthesia induction and maintenance will follow a TCI protocol with propofol and sufentanil, targeting a PSI between 30-50. The goal is rSO2 at or above 85% of baseline. If rSO2 drops below, a DO2 optimisation protocol will be activated, confirming anaesthetic depth and SpO2 levels. If SVV exceeds 12%, a 250 ml crystalloid bolus will be administered until SVV decreases. If SVRI is below 1600 dynes·s·m²/cm⁵, a norepinephrine bolus will be administered. CI will be monitored, and dobutamine will start if CI drops below 2.4 L/min/m². If rSO2 still remains low , head position, FIO2 and PEEP changes will be made.
  Interventions: Device: Multimodal monitoring
- Control (No Intervention): Sufentanil and propofol TCI dosing will be administered using Gepts and Schnider effect-site models, respectively. The anaesthesiologist will monitor the effect-site concentration of propofol during induction, titrating until the loss of eyelash reflex and response to verbal stimuli occur. The dose will then be increased by 20% and maintained until surgery completion. Following intubation, 0.03 mg/kg of midazolam will be given to ensure amnesia in case of inadvertent awareness. If the patient's HR or MAP increases by more than 20% above preoperative values, the propofol concentration will be increased by 0.3 mcg/ml. If intraoperative awareness is suspected, indicated by lacrimation or spontaneous respiration, an additional 0.03 mg/kg midazolam and 0.2 mg/kg esketamine will be administered. Rocuronium bromide will be given at 0.6 mg/kg LBW for intubation. Dosing of intravenous fluids, blood transfusions, vasopressors, and inotropes will be managed by the attending anaesthesiologist.

INTERVENTIONS:
Device: Multimodal monitoring — The rSO2 will be maintained during surgery by ensuring appropriate haemoglobin concentration and DO2 at or above 85% of baseline. If rSO2 falls below this level, a DO2 optimisation protocol will be activated, confirming anaesthetic depth and maintaining SpO2 levels. If SVV exceeds 12%, a crystalloid bolus of 250 ml will be administered until SVV decreases or no further increases in SVI occur. Should SVV be below 12%, the PPV to SVV ratio will be assessed, with continued crystalloid administration warranted for a ratio over 0.7. SVRI will be evaluated, and if SVRI is below 1600 dynes·s·m²/cm⁵, a norepinephrine bolus will be administered. A noticeable increase in MAP (>10%) will require a norepinephrine infusion to maintain MAP above 65 mmHg. If these measures do not suffice, CI will be monitored, and dobutamine will be infused if CI drops below 2.4 L/min/m². If rSO2 remains low after all interventions, adjustments to head position and increases in FiO2 or PEEP will be made.
  Arms: Interventional

SUMMARY:
This study will include patients aged 50 and older scheduled for elective abdominal oncologic surgery, classified as ASA II and III due to increased anaesthetic and surgical risk. Gender will not be a stratification factor. Exclusion criteria include patient refusal, memory impairment, psychosis, known or suspected EEG abnormalities, chronic psychoactive medication use, urgent procedures, BMI below 18 kg/m² or above 35 kg/m², persistent arrhythmias, NYHA class III-IV heart failure, valvular disease, liver diseases, and anticipated surgery duration over six hours. Eligible patients must sign an informed consent form one day prior to surgery. Demographic data collected will include age, sex, operation type, comorbidities, ASA status, height, weight, and BMI. Randomisation will occur before the study begins with a sample size of 100 subjects based on a pilot study of 5 patients per group.

Premedication and Monitoring: Patients will receive premedication per institutional protocol, which includes intramuscular midazolam. Intraoperative monitoring follows randomisation allocation. The control group will have standard measurements, including invasive pressure and ECG. Data collection will be handled by designated team members who will archive anaesthesia charts. After intubation, patients will be ventilated with 6-8 ml/kg of predicted body weight and a fresh gas flow of 1 L/min.

Intervention Group Protocol: In the intervention group, monitoring will be established via radial artery cannulation under local anaesthesia, using LiDCOrapid®, Rainbow®, and Hb attachments. Baseline MAP and CO values will be recorded, with DO2 calculated automatically. Sensors will be positioned to monitor anaesthetic depth and rSO2 before pre-oxygenation. A noradrenaline infusion will maintain venous tone.

Anaesthesia will use TCI with propofol and sufentanil, targeting specific values based on age groups. The primary goal is to maintain an rSO2 of at least 85% of baseline. If rSO2 falls below this threshold, a DO2 optimisation protocol will be initiated, adjusting conditions and administering fluids and medications as necessary.

Control Group Protocol: In the control group, propofol and sufentanil will be administered as previously outlined with adjustments based on intraoperative responses and awareness. Rocuronium bromide will be used for neuromuscular blockade, with monitoring and administration of fluids managed by the attending anaesthesiologist.

Data Recording: All data during procedures will be recorded digitally or manually, and post-procedure data will be downloaded for analysis. Patients will be transferred to the ICU for postoperative monitoring.

Laboratory Analysis: Blood samples for routine analysis will be collected at three time points: prior to surgery, upon ICU admission, and 24 hours after. Parameters assessed include complete blood count, electrolyte levels, PT, aPTT, fibrinogen, blood gas parameters, lactate, troponin I, and NTproBNP.

Outcome Measurements: Both groups will be monitored for duration of anaesthesia, drug administration, fluid volume, postoperative complications, mortality rates, and ICU length of stay (LOS). Continuous variables will be reported using descriptive statistics or interquartile ranges, while categorical variables will be shown as counts and percentages.

Statistical analysis will be performed using Mann Whitney U test for continuous variables, repeated measures ANOVA for group comparisons, and chi-squared tests for categorical variables. ANCOVA will be employed to compare clinical outcomes with age as a covariate. The software package jamovi v2.5.3 will be utilized for statistical analysis with a significance level set at p < 0.05.

DETAILED DESCRIPTION:
This study will include patients aged 50 years or older who are scheduled for elective abdominal oncologic surgery, specifically those classified as ASA II and ASA III due to their elevated anaesthetic and surgical risk profiles. Sex distribution will not serve as a stratification variable. Exclusion criteria encompass patient refusal; cognitive impairment; psychosis; known or suspected electroencephalographic disorders (including epilepsy or prior neurosurgical procedures); chronic use of psychoactive medications; urgent or emergent surgeries; body mass index (BMI) less than 18 kg/m² or greater than 35 kg/m²; persistent arrhythmias, including atrial fibrillation and undulation; documented NYHA class III-IV heart failure or preoperative left ventricular ejection fraction below 30%; significant valvular disease involving aortic or mitral stenosis or regurgitation; liver conditions such as decompensated cirrhosis and coagulopathies; and anticipated operative duration exceeding six hours. Eligible participants must provide written informed consent one day preceding surgery. Demographic information for both intervention and control groups will include age, sex, planned procedure type, comorbidities, ASA classification, height, weight, and BMI. Randomisation will be conducted prior to study initiation using https://www.random.org/ with a total sample size of 100 subjects. A pilot study was performed involving five patients in each group to inform sample size calculations.

Premedication will be administered to all patients according to institutional protocol and consists of intramuscular midazolam, with optional addition of atropine. Intraoperative monitoring will follow randomisation assignments. The control group will receive standard monitoring, including invasive pressure measurements, ECG, SpO2, IBP, and, when indicated, central venous pressure. Designated team members are responsible for data collection and archiving copies of the anaesthesia chart. In both groups, following intubation, patients will be connected to an anaesthesia machine (Dräger Perseus, Drägerwerk AG & Co. KGaA, Lübeck, Germany) and ventilated at 6-8 ml/kg of predicted body weight. Fresh gas flow will be maintained at 1 L/min, with FiO2 adjusted to ensure expiratory oxygen concentration remains between 30-40%. Upon completion of surgery, the attending anaesthesiologist will determine whether to continue mechanical ventilation and administer antidotes based on clinical judgement.

In the intervention group, patients will be monitored through radial artery cannulation performed under local anesthesia before induction. Monitoring devices used include LiDCOrapid®, Rainbow®, and an Hb module connected to the Root® monitor. Baseline measurements for mean arterial pressure (MAP) and cardiac output (CO) will be taken, with oxygen delivery (DO2) automatically calculated from the baseline CO and hemoglobin values detected by the Masimo Rainbow sensor. Prior to pre-oxygenation, SedLine® and O3® adult sensors will be attached to the patient's forehead to measure anaesthetic depth and regional oxygen saturation (rSO2), respectively. A low-dose infusion of noradrenaline (Noradrenalin Ligula Pharma, Laboratorios Normon S.A., Madrid, Spain; 1mg/50ml at 5 ml·hr-¹) will be started to help maintain venous tone.

Anaesthesia will be both induced and maintained using a target-controlled infusion (TCI) method with propofol (Propofol MCT Fresenius, Fresenius Kabi, Graz, Austria) and sufentanil (Sufentanil Altamedics, Altamedics GmbH, Cologne, Germany), delivered via the Braun Perfusor® Space system (B. Braun SE, Melsungen, Germany). The goal is to keep SedLine® values within a range of 30 to 50. Sufentanil dosing for intravenous induction will follow the Gepts effect-site model: for patients under 68 years, concentrations will be 0.5 ng/ml for induction, 0.3 ng/ml for maintenance, and 0.25 ng/ml for extubation. For those aged 69-79 years, the protocol calls for 0.35 ng/ml during induction, 0.25 ng/ml during maintenance, and 0.20 ng/ml at extubation. Patients over 79 years will receive 0.30 ng/ml for induction, 0.20 ng/ml for maintenance, and 0.17 ng/ml for extubation. Propofol will be administered according to the Schnider model, with 3 mcg/mL used for induction and 2-3 mcg/mL for maintenance.

The primary objective is to maintain rSO2 by ensuring adequate haemoglobin concentration and DO2 at or above 85% of baseline. Should rSO2 fall below this threshold, the at-tending anaesthesiologist will implement a DO2 optimization protocol: con-firming adequate anaesthetic depth, maintaining SpO2, and administering a 250 ml crystalloid bolus if stroke volume variation (SVV) exceeds 12%, repeated as needed until SVV drops below 12% or no further increase in stroke volume index (SVI) occurs. When SVV is below 12%, the PPV to SVV ratio will be assessed; if >0.7, crystalloid boluses will continue. Otherwise, systemic vascular resistance index (SVRI) will be evaluated, and a norepinephrine bolus (2-10 mcg) administered if SVRI is less than 1600 dynes·s·m²/cm⁵. If a significant MAP increase (>10%) follows, a norepinephrine infusion will be started and titrated to maintain MAP >65 mmHg. If not, the CI will be observed, and dobutamine infusion (Dobutamin Panpharma, Panpharma, Luitré, France) commenced if CI is below 2.4 L/min/m². If all measures fail to optimize rSO2, head position adjustments and increases in FiO2 and/or PEEP will be made until adequate rSO2 is achieved. For hypertension (systolic BP >180 mmHg) during appropriate anaesthetic depth, noradrenaline infusion will be discontinued. Maintenance fluids will be administered as balanced crystalloid (Iono-lyte, Fresenius Kabi Deutschland GmbH, Friedberg, Germany) at 4 mL/kg/h, aiming for urine output (UO) ≥0.5 mL/kg/h. Neuromuscular blockade will be achieved using rocu-ronium bromide (Esmeron, Merck Sharp & Dohme B.V., Haarlem, Netherlands) at 0.6 mg/kg lean body weight (LBW) for intubation and maintained with 6 mcg/kg/min LBW. At the conclusion of surgery, neuromuscular blockade will be reversed with sugammadex (Sugammadex Mylan, Mylan Pharmaceuticals Ltd., Dublin, Ireland).

Control group patients Sufentanil and propofol target-controlled infusion (TCI) dosing will be administered according to established protocols. The anaesthesiologist will monitor the effect-site concentration (Ce) of propofol during induction, adjusting the dosage until loss of eyelash reflex, absence of response to verbal stimuli, and onset of apnoea are observed; subsequently, Ce will be increased by 20% and maintained throughout the duration of surgery. Following intubation, 0.03 mg/kg midazolam (Midazolam Hameln, Hameln, Germany) will be administered to ensure amnesia in case of inadvertent awareness. If the patient's heart rate or mean blood pressure exceeds preoperative values by more than 20%, the propofol Ce will be increased by 0.3 mcg/ml. Signs suggestive of intraoperative awareness-including lacrimation, sweating, limb movement, or spontaneous respiration-will prompt administration of an additional 0.03 mg/kg midazolam and 0.2 mg/kg esketamine (Esgamda, G.L. Pharma GmbH, Lannach, Austria). Rocuronium bromide will be given at 0.6 mg/kg lean body weight for intubation, with supplemental 10 mg doses provided as necessary based on inadequate muscle relaxation (propofol Ce > 4.5 mcg/ml, as determined by the surgeon). Intravenous fluids (crystalloids and colloids), blood transfusions, vasopressors, and inotropes will be managed at the discretion of the attending anaesthesiologist.

Data Recording Masimo Root® monitors equipped with LiDCO®, Hb module, Sedline®, and O3® will be employed for the intervention group. All relevant data-including times of induction, incision, and intraoperative remarks-will be documented either on the Root® monitor or recorded separately when appropriate. Upon completion of each procedure, data will be extracted using Trace® software for the Root® system. As the anaesthesia record is maintained in a non-digital format, copies of the anaesthesia sheet containing all essential details must be produced and submitted together with the corresponding digital records. Following surgery, patients will be transferred to the ICU.

Laboratory Analysis Blood samples for routine laboratory investigations will be collected at three specific time points: prior to surgery, upon ICU admission, and 24 hours post-admission. Analyses will include complete blood count, electrolyte assessment, prothrombin time (PT), activated partial thromboplastin time (aPTT), fibrinogen concentration, blood gas parameters, lactate concentration, troponin I, and N-terminal pro-brain natriuretic peptide (NTproBNP).

The same parameters will be systematically monitored for both the control and intervention groups. Monitored variables include duration of anaesthesia (in minutes), administered medications, volume and type of infusions, quantity and type of blood components, intraoperative urine output, ICU length of stay, duration of mechanical ventilation, incidence of significant postoperative complications (e.g., cardiovascular events, acute kidney injury, cerebrovascular events), frequency of postoperative surgical complications (including re-operations), mortality rates at 7 and 30 days, as well as overall hospital length of stay.

Continuous variables are presented as either mean and standard deviation (SD) for descriptive statistics, or median and interquartile range (tables), and mean with 95% confidence interval (graphs) for inferential analysis. Normality of distribution was assessed using the Shapiro-Wilk test. Categorical variables are reported as counts and percentages.

Statistical significance of differences in continuous variables was evaluated using the Mann-Whitney U test, while repeated measurements between groups were analysed via repeated measures analysis of variance (RM-ANOVA) with post-hoc Holm-Šidák correction. Differences in categorical variables between groups were assessed using the chi-squared test or Fisher's exact test, as appropriate.

Analysis of covariance (ANCOVA), incorporating patient age as a covariate, was employed to compare clinical outcomes between groups. All statistical analyses, power calculations, and data visualizations were performed using the jamovi software package version 2.5.3. A p-value less than 0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* aged 50 years or older
* scheduled for elective major abdominal surgery, specifically those classified as ASA II and ASA III

Exclusion Criteria:

* patient refusal;
* memory impairment (psychosis);
* known or suspected electroencephalo-graphic abnormalities (such as epilepsy or previous brain surgery);
* chronic use of psy-choactive medication;
* urgent or emergent procedures;
* body mass index (BMI) below 18 kg/m2 or above 35 kg/m2;
* persistent arrhythmias including atrial fibrillation and undulation;
* documented NYHA class III-IV heart failure or a preoperative left ventricular ejection fraction below 30%;
* valvular disease involving aortic and/or mitral stenosis or regurgita-tion;
* liver diseases such as decompensated cirrhosis and coagulopathies;
* anticipated operation duration exceeding six hours.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Duration of mechanical ventilation | From enrollment to the end of treatment at 30 days
  Patients in the Interventional group should have shorter duration of mechanical ventilation after surgery

SECONDARY OUTCOMES:
troponin I levels | From enrollment to the end of treatment at 30 days
  Patients in the Interventional group should have lower levels of troponin I upon admission to the ICU, and 24 hours post-admission, a lower rise in that value compared to preoperative value
NTproBNP levels | From enrollment to the end of treatment at 30 days
  Patients in the Interventional group should have lower levels of N-terminal brain natriuretic peptide upon admission to the ICU, and 24 hours post-admission, a lower rise in that value compared to preoperative value
Lactate levels | From enrollment to the end of treatment at 30 days
  Patients in the Interventional group should have lower levels of lactate upon admission to the ICU, and 24 hours post-admission, a lower rise in that value compared to preoperative value
postoperative medical complications | From enrollment to the end of treatment at 30 days
  Patients in the Interventional group should have lower incidence of significant postoperative complications (such as cardiovascular events, acute kidney injury, or cerebrovascular events)
post-operative surgical complications | From enrollment to the end of treatment at 30 days
  Patients in the Interventional group should have lower frequency of post-operative surgical complications (including re-operation)
ICU LOS | From enrollment to the end of treatment at 30 days
  Patients in the Interventional group should have shorter lenght of stay in the intensive care unit
Mortality 7 days | From enrollment to the end of treatment at 30 days
  Patients in the Interventional group should have smaller mortality rate at 7 days after surgery
Mortality 30 days | From enrollment to the end of treatment at 30 days
  Patients in the Interventional group should have smaller mortality rate at 30 days after surgery
Hospital LOS | From enrollment to the end of treatment at 30 days
  The patients in the interventional group shold have shorter hospital lenght of stay

CONTACTS AND LOCATIONS:
Overall Officials: Jasminka Peršec, M.D., PhD, Ass. Prof, Study Chair — University Hospital Dubrava; Andrej Šribar, Assoc. Prof., MD, PhD, Study Chair — University Hospital Dubrava
Locations (1):
- University hospital Dubrava, Zagreb, Croatia, Croatia

IPD SHARING:
Plan to Share IPD: Yes
All data are available, and will remain accessible, in Microsoft Excel format in both anonymous and coded versions following a written request to the authors.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: From June 1st, 2026 until December 31st, 2027
Access Criteria: Individuals who submit a formal, written request will have their submissions evaluated by the Study Group, and permission will be granted accordingly.

REFERENCES:
- [Background] Silva-Jr JM, Menezes PFL, Lobo SM, de Carvalho FHS, de Oliveira MAN, Cardoso Filho FNF, Fernando BN, Carmona MJC, Teich VD, Malbouisson LMS. Impact of perioperative hemodynamic optimization therapies in surgical patients: economic study and meta-analysis. BMC Anesthesiol. 2020 Mar 31;20(1):71. doi: 10.1186/s12871-020-00987-y. PMID 32234025
- [Background] Sadique Z, Harrison DA, Grieve R, Rowan KM, Pearse RM; OPTIMISE study group. Cost-effectiveness of a cardiac output-guided haemodynamic therapy algorithm in high-risk patients undergoing major gastrointestinal surgery. Perioper Med (Lond). 2015 Dec 14;4:13. doi: 10.1186/s13741-015-0024-x. eCollection 2015. PMID 26674494
- [Background] Kouz K, Bergholz A, Diener O, Leistenschneider M, Thompson C, Pichotka F, Trepte C, Schwedhelm E, Renne T, Krause L, Nicklas JY, Saugel B. Effect of intraoperative personalized goal-directed hemodynamic management on acute myocardial injury in high-risk patients having major abdominal surgery: a post-hoc secondary analysis of a randomized clinical trial. J Clin Monit Comput. 2022 Dec;36(6):1775-1783. doi: 10.1007/s10877-022-00826-0. Epub 2022 Feb 24. PMID 35201549
- [Background] Moharari RS, Shahinpour S, Etezadi F, Najafi A, Khajavi MR, Pourfakhr P. Comparison of Goal-Directed Fluid Therapy using LiDCOrapid System with Regular Fluid Therapy in Patients Undergoing Spine Surgery as a Randomised Clinical Trial. Rom J Anaesth Intensive Care. 2022 Sep 25;28(1):1-9. doi: 10.2478/rjaic-2021-0001. eCollection 2021 Jul. PMID 36846537
- [Background] Tengberg LT, Bay-Nielsen M, Bisgaard T, Cihoric M, Lauritsen ML, Foss NB; AHA study group. Multidisciplinary perioperative protocol in patients undergoing acute high-risk abdominal surgery. Br J Surg. 2017 Mar;104(4):463-471. doi: 10.1002/bjs.10427. Epub 2017 Jan 23. PMID 28112798
- [Background] Vignon P, Evrard B, Asfar P, Busana M, Calfee CS, Coppola S, Demiselle J, Geri G, Jozwiak M, Martin GS, Gattinoni L, Chiumello D. Fluid administration and monitoring in ARDS: which management? Intensive Care Med. 2020 Dec;46(12):2252-2264. doi: 10.1007/s00134-020-06310-0. Epub 2020 Nov 9. PMID 33169217
- [Background] Gurgel ST, do Nascimento P Jr. Maintaining tissue perfusion in high-risk surgical patients: a systematic review of randomized clinical trials. Anesth Analg. 2011 Jun;112(6):1384-91. doi: 10.1213/ANE.0b013e3182055384. Epub 2010 Dec 14. PMID 21156979
- [Background] Thomsen KK, Sessler DI, Krause L, Hoppe P, Opitz B, Kessler T, Chindris V, Bergholz A, Flick M, Kouz K, Zollner C, Schulte-Uentrop L, Saugel B. Processed electroencephalography-guided general anesthesia and norepinephrine requirements: A randomized trial in patients having vascular surgery. J Clin Anesth. 2024 Aug;95:111459. doi: 10.1016/j.jclinane.2024.111459. Epub 2024 Apr 9. PMID 38599161
- [Background] Huang L, Liu LL, Lu YD, Zhuang MY, Dou W, Liu H, Ji FH, Peng K. Assessing Sedation Depth with PSI in Elderly ERCP Patients: A Prospective Cohort Study. Clin Interv Aging. 2025 Feb 11;20:137-145. doi: 10.2147/CIA.S504212. eCollection 2025. PMID 39959307
- [Background] Green DW. A retrospective study of changes in cerebral oxygenation using a cerebral oximeter in older patients undergoing prolonged major abdominal surgery. Eur J Anaesthesiol. 2007 Mar;24(3):230-4. doi: 10.1017/S0265021506001645. Epub 2006 Oct 23. PMID 17054814
- [Background] Green D, Bidd H, Rashid H. Multimodal intraoperative monitoring: an observational case series in high risk patients undergoing major peripheral vascular surgery. Int J Surg. 2014;12(3):231-6. doi: 10.1016/j.ijsu.2013.12.016. Epub 2014 Jan 8. PMID 24412536
- [Background] Yue C, Su L, Wang J, Cui N, Zhou Y, Cheng W, Tang B, Rui X, He H, Long Y. Prediction of mechanical ventilation outcome by early abdominal-visceral-blood-flow-and-function score in critically ill patients after cardiopulmonary bypass in the ICU: A prospective observational study. J Intensive Med. 2023 Oct 18;4(1):101-107. doi: 10.1016/j.jointm.2023.09.001. eCollection 2024 Jan. PMID 38263967
- [Background] Clark MG, Mueller DA, Dudaryk R, Li G, Freundlich RE. Patient and Operative Factors Predict Risk of Discretionary Prolonged Postoperative Mechanical Ventilation in a Broad Surgical Cohort. Anesth Analg. 2023 Mar 1;136(3):524-531. doi: 10.1213/ANE.0000000000006205. Epub 2022 Oct 13. PMID 36634028
- [Background] Murthy SC, Arroliga AC, Walts PA, Feng J, Yared JP, Lytle BW, Blackstone EH. Ventilatory dependency after cardiovascular surgery. J Thorac Cardiovasc Surg. 2007 Aug;134(2):484-90. doi: 10.1016/j.jtcvs.2007.03.006. PMID 17662794
- [Background] Qiu L, Ma Y, Ge L, Zhou H, Jia W. Efficacy of Cerebral Oxygen Saturation Monitoring for Perioperative Neurocognitive Disorder in Adult Noncardiac Surgical Patients: A Systematic Review and Meta-Analysis of Randomized Controlled Trials. World Neurosurg. 2025 Feb;194:123570. doi: 10.1016/j.wneu.2024.123570. Epub 2025 Jan 23. PMID 39701521
- [Background] Ding L, Chen DX, Li Q. Effects of electroencephalography and regional cerebral oxygen saturation monitoring on perioperative neurocognitive disorders: a systematic review and meta-analysis. BMC Anesthesiol. 2020 Sep 30;20(1):254. doi: 10.1186/s12871-020-01163-y. PMID 32998697
- [Background] Staicu RE, Vernic C, Ciurescu S, Lascu A, Aburel OM, Deutsch P, Rosca EC. Postoperative Delirium and Cognitive Dysfunction After Cardiac Surgery: The Role of Inflammation and Clinical Risk Factors. Diagnostics (Basel). 2025 Mar 26;15(7):844. doi: 10.3390/diagnostics15070844. PMID 40218194
- [Background] Wang X, Feng K, Liu H, Liu Y, Ye M, Zhao G, Wang T. Regional cerebral oxygen saturation and postoperative delirium in endovascular surgery: a prospective cohort study. Trials. 2019 Aug 14;20(1):504. doi: 10.1186/s13063-019-3586-y. PMID 31412906
- [Background] Tang L, Kazan R, Taddei R, Zaouter C, Cyr S, Hemmerling TM. Reduced cerebral oxygen saturation during thoracic surgery predicts early postoperative cognitive dysfunction. Br J Anaesth. 2012 Apr;108(4):623-9. doi: 10.1093/bja/aer501. Epub 2012 Feb 5. PMID 22311364
- [Background] Zhang CY, Yang YS, Pei MQ, Chen XL, Chen WC, He HF. The Association of Cerebral Oxygen Desaturation with Postoperative Cognitive Dysfunction in Older Patients: A Review. Clin Interv Aging. 2024 Jun 17;19:1067-1078. doi: 10.2147/CIA.S462471. eCollection 2024. PMID 38911674
- [Background] Murkin JM, Adams SJ, Novick RJ, Quantz M, Bainbridge D, Iglesias I, Cleland A, Schaefer B, Irwin B, Fox S. Monitoring brain oxygen saturation during coronary bypass surgery: a randomized, prospective study. Anesth Analg. 2007 Jan;104(1):51-8. doi: 10.1213/01.ane.0000246814.29362.f4. PMID 17179242
- [Background] Sala F, Niimi Y, Berenstein A, Deletis V. Role of Multimodality Intraoperative Neurophysiological Monitoring during Embolisation of a Spinal Cord Arteriovenous Malformation. A Paradigmatic Case. Interv Neuroradiol. 2000 Sep 30;6(3):223-34. doi: 10.1177/159101990000600308. Epub 2001 May 15. PMID 20667201
- [Background] Linton NW, Linton RA. Estimation of changes in cardiac output from the arterial blood pressure waveform in the upper limb. Br J Anaesth. 2001 Apr;86(4):486-96. doi: 10.1093/bja/86.4.486. PMID 11573621
- [Background] De Keijzer IN, Massari D, Niezen CK, Bokkers RPH, Vos JJ, Scheeren TWL. Agreement of somatic and renal near-infrared spectroscopy with reference blood samples during a controlled hypoxia sequence: a healthy volunteer study. J Clin Monit Comput. 2023 Jun;37(3):805-814. doi: 10.1007/s10877-022-00944-9. Epub 2022 Dec 4. PMID 36463540
- [Background] Drover D, Ortega HR. Patient state index. Best Pract Res Clin Anaesthesiol. 2006 Mar;20(1):121-8. doi: 10.1016/j.bpa.2005.07.008. PMID 16634419
- [Background] Green DW, Kunst G. Cerebral oximetry and its role in adult cardiac, non-cardiac surgery and resuscitation from cardiac arrest. Anaesthesia. 2017 Jan;72 Suppl 1:48-57. doi: 10.1111/anae.13740. PMID 28044331
- [Background] Salzwedel C, Puig J, Carstens A, Bein B, Molnar Z, Kiss K, Hussain A, Belda J, Kirov MY, Sakka SG, Reuter DA. Perioperative goal-directed hemodynamic therapy based on radial arterial pulse pressure variation and continuous cardiac index trending reduces postoperative complications after major abdominal surgery: a multi-center, prospective, randomized study. Crit Care. 2013 Sep 8;17(5):R191. doi: 10.1186/cc12885. PMID 24010849
- [Background] Shoemaker WC, Appel PL, Kram HB, Waxman K, Lee TS. Prospective trial of supranormal values of survivors as therapeutic goals in high-risk surgical patients. Chest. 1988 Dec;94(6):1176-86. doi: 10.1378/chest.94.6.1176. PMID 3191758
- [Background] Dobson GR, Chau A, Denomme J, Frost S, Fuda G, Mc Donnell C, Milkovich R, Milne AD, Sparrow K, Subramani Y, Young C. Guidelines to the Practice of Anesthesia-Revised Edition 2025. Can J Anaesth. 2025 Jan;72(1):15-63. doi: 10.1007/s12630-024-02906-y. Epub 2025 Feb 3. PMID 39900856
- [Background] Zajak J, Paral J, Sirovy M, Odlozilova S, Vinklerova K, Balik M, Cecka F. Methods of Blood Loss Quantification in Major Abdominal Surgery: A Narrative Review. Acta Medica (Hradec Kralove). 2023;66(4):133-137. doi: 10.14712/18059694.2024.7. PMID 38588390
- [Background] Myles PS, Bellomo R, Corcoran T, Forbes A, Peyton P, Story D, Christophi C, Leslie K, McGuinness S, Parke R, Serpell J, Chan MTV, Painter T, McCluskey S, Minto G, Wallace S; Australian and New Zealand College of Anaesthetists Clinical Trials Network and the Australian and New Zealand Intensive Care Society Clinical Trials Group. Restrictive versus Liberal Fluid Therapy for Major Abdominal Surgery. N Engl J Med. 2018 Jun 14;378(24):2263-2274. doi: 10.1056/NEJMoa1801601. Epub 2018 May 9. PMID 29742967
- See also: LiDCOrapid. LiDCO - Hemodynamic Monitoring for the entire patient pathway — https://www.lidco.com/product/lidco-rapid
- See also: 17. jamovi - open statistical software for the desktop and cloud — https://www.jamovi.org